CLINICAL TRIAL: NCT00803010
Title: Phase II Trial of Tacrolimus and Rapamycin vs. Tacrolimus and Methotrexate as GVHD Prophylaxis After Allogeneic Peripheral Blood Hematopoietic Cell Transplantation
Brief Title: Graft-Versus-Host Disease (GVHD) Prophylaxis After Allogeneic Peripheral Blood Hematopoietic Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCC-15372; IRB 106591
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2013-12

CONDITIONS: Acute Graft Versus Host Disease
Keywords: Acute Graft Versus Host Disease (aGVHD); GVHD; graft-versus-host disease; tacrolimus; sirolimus; methotrexate; combination therapy; GVHD prophylaxis
MeSH Terms: conditions — Graft vs Host Disease | interventions — Tacrolimus; Methotrexate; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrolimus / Rapamycin (TAC/RAPA) (Active Comparator): Tacrolimus: beginning 3 days before transplant and given for at least 50 days.
  Rapamycin: given the day before transplant and continued daily for at least one year.
  Interventions: Drug: Tacrolimus (TAC); Drug: Rapamycin (RAPA)
- Tacrolimus / Methotrexate (TAC/MTX) (Active Comparator): Tacrolimus: beginning 3 days before transplant and given for at least 50 days.
  Methotrexate: given on days 1, 3, 6 and 11, after transplant.
  Interventions: Drug: Tacrolimus (TAC); Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: Tacrolimus (TAC) — Tacrolimus: administered at 0.02 mg/kg/day (based on ideal body weight) continuous IV infusion or equivalent oral dosing starting on day -3.
  Other Names: FK-506; fujimycin; Prograf; Advagraf; Protopic
Drug: Methotrexate (MTX) — Methotrexate: administered on day 1 at dose of 15 mg/m^2, and a dose of 10 mg/m^2 on days 3, 6, and 11. Dose can be adjusted for reduced creatinine clearance.
  Other Names: Trexall; Rheumatrex
  Arms: Tacrolimus / Methotrexate (TAC/MTX)
Drug: Rapamycin (RAPA) — Rapamycin: initially as 9 mg oral loading dose on day -1. Thereafter, administered as an oral regimen of 4 mg daily.
  Other Names: Sirolimus
  Arms: Tacrolimus / Rapamycin (TAC/RAPA)

SUMMARY:
The purpose of this research is to compare the effectiveness of Tacrolimus and Rapamycin to Tacrolimus and Methotrexate in the prevention of severe graft-versus-host-disease. Graft-versus-host-disease (GVHD) is a risk associated with allogeneic hematopoietic cell transplants (HCT). An allogeneic hematopoietic cell transplant is a transplant using bone marrow and blood cells that come from someone other than the patient (a donor).

DETAILED DESCRIPTION:
All drugs used in this study have been used in the prevention of graft-versus-host-disease after allogeneic hematopoietic cell transplant. Tacrolimus and Methotrexate used in combination are currently used as standard of care in the prevention of graft-versus-host-disease after allogeneic hematopoietic cell transplant. Tacrolimus and Rapamycin is a newer combination we are testing to see if it would be better than Tacrolimus and Methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 and ≤ 70
* Signed informed consent
* Adequate vital organ function
* No active infection, or asymptomatic infection well controlled by antibiotic HIV negative by ELISA or RT-PCR [if ELISA is positive and RT-PCR is negative, the ELISA is considered false positive]
* Hepatitis B and C negative by serology or RT-PCR
* Performance status: Karnofsky Performance Status Score ≥ 60%.

Exclusion Criteria:

* Those with any Sorror's co-morbidity factors with score > 3
* 2 or more Sorror's factors with composite score of ≥ 3

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Anasetti, MD, Study Director — HLeeMoffittCancerCenter
Locations (1):
- H.Lee Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- [Derived] Pidala J, Kim J, Jim H, Kharfan-Dabaja MA, Nishihori T, Fernandez HF, Tomblyn M, Perez L, Perkins J, Xu M, Janssen WE, Veerapathran A, Betts BC, Locke FL, Ayala E, Field T, Ochoa L, Alsina M, Anasetti C. A randomized phase II study to evaluate tacrolimus in combination with sirolimus or methotrexate after allogeneic hematopoietic cell transplantation. Haematologica. 2012 Dec;97(12):1882-9. doi: 10.3324/haematol.2012.067140. Epub 2012 Jun 11. PMID 22689677
- See also: H.Lee Moffitt Cancer Center & Research Institute — http://www.moffitt.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited between 09/10/2008 through 05/13/2011 from the Blood and Marrow Transplant Program patient population.
Groups:
- 1 Tacrolimus / Rapamycin: Tacrolimus / Rapamycin
  Tacrolimus and Rapamycin (Sirolimus): Tacrolimus - 0.02 mg/kg/day (based on ideal body weight) continuous IV infusion or equivalent oral dosing starting on day -3.
  Rapamycin - initially as 9 mg oral loading dose on day -1. Thereafter, administered as an oral regimen of 4 mg daily.
- 2 Tacrolimus / Methotrexate: Tacrolimus / Methotrexate
  Tacrolimus and Methotrexate: Tacrolimus administered at 0.02 mg/kg/day (based on ideal body weight) continuous IV infusion or equivalent oral dosing starting on day -3
  Methotrexate: administered on day 1 at dose of 15 mg/m^2, and a dose of 10 mg/m^2 on days 3, 6, and 11. Dose can be adjusted for reduced creatinine clearance.
Period: Overall Study
Arm/Group | 1 Tacrolimus / Rapamycin | 2 Tacrolimus / Methotrexate
Started | 37 | 37
Completed | 37 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Based on our preliminary data collected from patients receiving TAC/MTX, the acute GVHD (aGVHD) rate is estimated to be 80% at 100 days. A two-sided log-rank test will achieve 90% power at a 0.1 significance level. The result of this calculation serves as an approximation of power/sample size for the test we propose to use for the primary endpoint.
Groups:
- Tacrolimus / Rapamycin: Tacrolimus / Rapamycin
  Tacrolimus / Rapamycin: Tacrolimus - 0.02 mg/kg/day (based on ideal body weight) continuous IV infusion or equivalent oral dosing starting on day -3.
  Rapamycin - initially as 9 mg oral loading dose on day -1. Thereafter, administered as an oral regimen of 4 mg daily.
- Tacrolimus / Methotrexate: Tacrolimus / Methotrexate
  Tacrolimus / Methotrexate: Tacrolimus administered at 0.02 mg/kg/day (based on ideal body weight) continuous IV infusion or equivalent oral dosing starting on day -3
  Methotrexate: administered on day 1 at dose of 15 mg/m^2, and a dose of 10 mg/m^2 on days 3, 6, and 11. Dose can be adjusted for reduced creatinine clearance.
- Total: Total of all reporting groups
Arm/Group | Tacrolimus / Rapamycin | Tacrolimus / Methotrexate | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Continuous [Median (Full Range); unit: years] | 49 [25 to 68] | 48 [23 to 69] | 49 [23 to 69]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 34 | 68
  >=65 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 28 | 23 | 51
Region of Enrollment [Number; unit: participants]
  United States | 37 | 37 | 74

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Evidence of Acute Graft Versus Host Disease (aGVHD), Post Transplant
Description: Incidence of acute graft versus host disease grades 2-3 according to the Common Toxicity Criteria (CTC) version 3.
  Graft-versus-host-disease (GVHD) is a risk associated with allogeneic hematopoietic cell transplants (HCT). Clinical evidence of acute GVHD was recorded per standard grading scheme.
  Acute GVHD classified as the following:
  1. classic acute GVHD - onset within 100 days after transplant
  2. persistent - acute GVHD with onset prior to day 100 and without resolution beyond day 100
  3. recurrent - acute GVHD recurrent after prior episode of acute GVHD
  4. late acute GVHD - syndrome consistent with acute GVHD, without features of chronic GVHD, with onset occurring beyond 100 days
Time Frame: 100 Days Post Transplant
Population: All participants who received treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 1 Tacrolimus / Rapamycin | 2 Tacrolimus / Methotrexate
Number analyzed (Participants) | 37 | 37
percentage of participants | 43 [27 to 59] | 89 [72 to 96]

2. Secondary Outcome: Incidence of Increased Absolute Numbers of Regulatory T Cells (Treg)
Description: Absolute numbers of Treg at designated time points according to study arm. MTX = methotrexate/tacrolimus-treated patients; SIR = sirolimus/tacrolimus-treated patients; Treg absolute number units = number of cells/microL. A two-sided Wilcoxon's rank-sum test was employed to test differences in percent Treg (% Treg/total CD4+ cells).
Time Frame: 30 days and 90 days
Measure: Median (95% Confidence Interval); unit: Cells/MicroL
Arm/Group | 1 Tacrolimus / Rapamycin | 2 Tacrolimus / Methotrexate
Number analyzed (Participants) | 37 | 37
Cells/MicroL
  30 Day Measure | 16.27 [12.49 to 17.89] | 9.87 [8.59 to 13.47]
  90 Day Measure | 14.6 [10.76 to 18.1] | 9.67 [7.48 to 11.56]

3. Secondary Outcome: 2 Year Post Transplant Overall Survival (OS) Rate
Description: Defined as time from transplantation (day 0 as day of stem cell infusion per standard nomenclature) to death from any cause .
Time Frame: 2 years
Population: All participants who received treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 1 Tacrolimus / Rapamycin | 2 Tacrolimus / Methotrexate
Number analyzed (Participants) | 37 | 37
percentage of participants | 61 [41 to 77] | 69 [48 to 83]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Tacrolimus / Rapamycin | Tacrolimus / Methotrexate
Serious Adverse Events (participants affected / at risk) | 3/37 | 2/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus / Rapamycin (N=37) | Tacrolimus / Methotrexate (N=37)
Cardiac General - Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) — Cardiac General - Pericardial effusion, Grade 3
Hemorrhage, GI-Lower GI NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatobiliary/Pancreas - Abdominal pain secondary to acute cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) — Hepatobiliary / Pancreas, Grade 3 Abdominal pain secondary to acute cholecystitis
Renal / Genitourinary - Obstruction, GU Bladder (Renal and urinary disorders) | 0 (0) | 1 (1) — Obstruction, GU Bladder Grade 3 Bilateral ureteral obstruction secondary to clots
Renal / Genitourinary - Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) — Renal Failure Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No